CLINICAL TRIAL: NCT04252573
Title: Prospective, Multicenter, Non-randomized Study With Consecutive, Eligible Subject Enrollment at Each Site, for the Evaluation of the ChEVAS System for Endovascular Repair of Paravisceral, Juxtarenal, and Pararenal Abdominal Aortic Aneurysms.
Brief Title: Chimney EndoVascular Aneurysm Sealing Of New Expanded Indication
Acronym: ChEVAS One
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Endologix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-0015
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-11

CONDITIONS: 1 Paravisceral Abdominal Aortic Aneurysm; 2 Juxtarenal Abdominal Aortic Aneurysm; 3 Pararenal Abdominal Aortic Aneurysm; 4 Complex Abdominal Aortic Aneurysms
Keywords: Paravisceral Abdominal Aortic Aneurysm; Juxtarenal Abdominal Aortic Aneurysm; Pararenal Abdominal Aortic Aneurysm; Complex Abdominal Aortic Aneurysm; Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- ChEVAS System (Experimental): The ChEVAS procedure involves the use of the Nellix System in conjunction with parallel branch chimney stents for the treatment of juxtarenal, pararenal, or paravisceral abdominal aortic aneurysms.
  Interventions: Device: Chimney Endovascular Aortic Sealing (ChEVAS) System

INTERVENTIONS:
Device: Chimney Endovascular Aortic Sealing (ChEVAS) System — The ChEVAS procedure involves the use of the Nellix System in conjunction with parallel branch chimney stents for the treatment of juxtarenal, pararenal, or paravisceral abdominal aortic aneurysms.
  Other Names: ChEVAS

SUMMARY:
Prospective, multi-center, non-randomized study with consecutive, eligible subject enrollment at each site, for the evaluation of the ChEVAS System for Endovascular Repair of Complex Abdominal Aortic Aneurysms.

DETAILED DESCRIPTION:
This is a prospective multicenter study with consecutive eligible subject enrollment at each site. Enrollment will include up to 150 subjects (120 ChEVAS subjects and up to 30 infrarenal roll-in subjects). The ChEVAS study will evaluate the safety and effectiveness outcomes following appropriate government and ethics committee/IRB requirements and guidelines.

All enrolled (ChEVAS and Infrarenal) subjects will undergo a high resolution, contrast-enhanced computed tomography angiography (CT) scan of the relevant aortic and aortoiliac vasculature within three months of the scheduled procedure and at specified follow-up intervals post-implantation. Follow-up visits will occur at 30-days, 6-months, and annually to 5-years to assess aneurysm morphology, the status of the implanted devices, and relevant laboratory test results.

*As of October 27, 2021 ChEVAS ONE Study is voluntarily closed to screening and consenting. 13 subjects enrolled in the study will continue to be observed through 5-years.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18-years old
* Subject provided informed consent
* Subject agrees to all follow-up visits
* Abdominal aortic aneurysm (AAA) with maximum sac diameter ≥5.0 cm, or ≥ 4.5 cm which has increased by ≥ 0.5cm within the last 6-months, or which exceeds 1.5 times the transverse dimension of an adjacent non-aneurysmal aortic segment. No AAA <4cm will be included
* Absence of significant cranial angulation of the visceral vessels that would preclude vessel cannulation and stenting

Exclusion Criteria:

* Requirement of home oxygen
* Psychiatric or other condition that may interfere with the study
* Participating in another clinical drug and/or device study, which could confound the results of this study (patient must have completed the primary endpoint of any previous study at least 30-days prior to enrollment in this study)
* Known allergy or contraindication to any device material, contrast, or anticoagulants
* Serum creatinine level >1.8mg/dL
* CVA or MI within three months of enrollment/treatment
* Prior stent in any target visceral vessel, the aorta or iliac artery that may interfere with delivery system introduction or stent placement
* Connective tissue diseases (e.g., Marfan Syndrome)
* Unsuitable vascular anatomy that may interfere with device introduction or deployment
* Pregnant, planning to become pregnant within 60 months, or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2028-03 (Estimated)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Valley Vascular Consultants, Huntsville, Alabama
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - St Vincent Medical Group, Indianapolis, Indiana
  - University of Missouri, Columbia, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Providence Portland, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ChEVAS System
Started | 13
Completed | 0
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | ChEVAS System
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 8
  Non-Caucasian | 5
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Technical Success, Safety and Effectiveness Indicators at One-Month Post-Index Procedure
Description: The outcome at one-month post index procedure will be measured by the proportion of subjects that experience technical success and the absence of severe bowel ischemia, permanent paraplegia/paraparesis, renal failure, disabling stroke, abdominal aortic aneurysm rupture, and aneurysm-related mortality within 30-days of the index procedure.
Time Frame: 1-Month
Measure: Count of Participants; unit: Participants
Arm/Group | ChEVAS System
Number analyzed (Participants) | 13
Participants | 13

2. Primary Outcome: Proportion of Safety and Effectiveness Indicators at One-Year Post-Index Procedure
Description: The outcome at one-year post index procedure will be measured by the proportion of subjects that experience freedom from abdominal aortic aneurysm rupture and aneurysm-related mortality up until 1-year (day 365), freedom from imaging-related findings in the 1-year window (Type 1 or 3 endoleak, migration > 10mm, AAA sac expansion > 5mm, and occlusion within the ChEVAS System not seen at the index procedure), and open conversion through day 365.
Time Frame: 1-Year
Measure: Count of Participants; unit: Participants
Arm/Group | ChEVAS System
Number analyzed (Participants) | 13
Participants | 10

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | ChEVAS System
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 4/13
Other Adverse Events (participants affected / at risk) | 6/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ChEVAS System (N=13)
Hypertension (Cardiac disorders) | 3 (3)
Compartment Syndrome (Surgical and medical procedures) | 1 (1)
Neurological (Nervous system disorders) | 2 (2)
Endoleak Type 1A (Vascular disorders) | 1 (1)
Miscellaneous- Inguinal hernia (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ChEVAS System (N=13)
Bleeding/Anemia (Surgical and medical procedures) | 1 (1)
Cardiac (Cardiac disorders) | 1 (1)
Miscellaneous (General disorders) | 1 (1)
Nellix Device (Product Issues) | 2 (2)
Surgical Site Wound (Surgical and medical procedures) | 1 (1)
Vascular (Vascular disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-13): https://cdn.clinicaltrials.gov/large-docs/73/NCT04252573/Prot_SAP_000.pdf